CLINICAL TRIAL: NCT03901846
Title: Duration of ColdZyme® II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymatica AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CI70
Record Dates: First submitted 2019-04-02; First posted 2019-04-03 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ColdZyme (Other): The study is intended to verify the method used to measure the duration of ColdZyme®.
  Each participant will be his own control as samples are taken before application of ColdZyme and used as an internal control.
  Interventions: Device: ColdZyme

INTERVENTIONS:
Device: ColdZyme — ColdZyme is a Class I medical device (CE-marked) with the following composition: glycerol, water, Tris buffer, CaCl2, menthol and trypsin

SUMMARY:
The objective of this investigation is to verify that ColdZyme® is deposited onto the throat and estimate the half-life of the ColdZyme® solution in the oropharynx of human volunteers using a log-linear mixed-effects model (LMM).

DETAILED DESCRIPTION:
The study is an Open Label, Non-Comparative study intended to verify the method used to measure the duration of ColdZyme®. Each participant will be his own control as samples are taken before application of ColdZyme and used as an internal control. Samples will be taken from the oropharyngeal membrane using a cotton swab before application, and 1, 3, 5, 10, 20, and 60 minutes after application. Glycerol will then be extracted from the swabs using water and the concentration of glycerol will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between 18-70 years. The investigator judges the definition of healthy by medical history.
* No reported symptoms of sore throat.
* Readiness to comply with trial procedures.
* Females of childbearing potential: should use reliable method of birth control.
* Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

* Known allergy or hypersensitivity to the components of the investigational product
* History and/or presence of clinically significant condition/disorder (self-reported), which per investigator's judgement could interfere with the results of the study or the safety of the subject.
* Any current cold symptom such as sore throat, sneezing, rhinorrhea, malaise, nasal obstruction or cough.
* Use of products, drugs, or food containing glycerol that may influence the study outcome, or concomitant medication with pharmaceuticals that might cause dry mouth (xerostomia), e.g. but not restricted to, morphine or morphine derivates, diuretics, antidepressants or other drugs with anticholinergic effect.
* Females: Pregnant or breast-feeding
* History of (in the past 12 months prior to study start) or current abuse of drugs, alcohol or medication
* Inability to comply with study requirements according to investigator's judgement
* Participation in another clinical study in the 30 days prior to enrolment and during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Duration of the ColdZyme barrier | 0-60 minutes
  To measure the duration of the ColdZyme barrier following intra-oral deposition, by analyzing the oro-pharyngeal glycerol amount over time between 0 and 60 minutes after application.

CONTACTS AND LOCATIONS:
Overall Officials: Bardur Sigurgeirsson, MD, PhD, Principal Investigator — Cutis Clinical Research Center (CCRC)
Locations (1):
- Cutis Clinical Research Center, Kopavogur, Iceland

IPD SHARING:
Plan to Share IPD: No